CLINICAL TRIAL: NCT00844025
Title: Pharmaceutical Care and Clinical Outcomes for the Elderly Taking Potentially Inappropriate Medication: a Randomized-Controlled Trial
Brief Title: Pharmaceutical Care and Clinical Outcomes for the Elderly Taking Potentially Inappropriate Medication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Tsai Ming Dar/Chief of Shin Kong Wu Ho-Su Memorial Hospital Research and Education Assessment Department, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SKH-8302-98-NDR-05
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Elderly; Chronic Disease
Keywords: Adverse drug reaction; Inappropriate medication; Pharmacist; Pharmaceutical care
MeSH Terms: conditions — Chronic Disease; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacist intervention (Experimental): Patients in the intervention group will receive pharmaceutical care delivered by clinical pharmacist, which including medication review, medication reconciliation, patient education and recommended actions.
  Interventions: Behavioral: Pharmacist intervention
- Usual care (No Intervention): Patients randomized to usual care group will receive routine review of medication by ward-based pharmacist and nurse.

INTERVENTIONS:
Behavioral: Pharmacist intervention — Medication review, medication reconciliation, and pharmacotherapy recommendation.
  Arms: Pharmacist intervention

SUMMARY:
The investigators propose that clinical pharmacist interventions would reduce the rate of adverse drug events in elderly patients taking potentially inappropriate medication.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients aged at least 65 years
* Taking at least six prescribed medicines regularly, including at least one potential inappropriate medication

Exclusion Criteria:

* Patients who refused informed consent
* Discharged before consent could be obtained
* Cognitive impaired

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Number of unsolved drug-related problems | 14 days after randomization

SECONDARY OUTCOMES:
Rate of adverse drug event during hospitalization | 14 days after randomization
Number of potentially inappropriate medication | 14 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Liu Jen Wei, MS, Principal Investigator — Shin Kong Wo Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wo Ho-Su Memorial Hospital, Department of Pharmacy, Taipei, Taiwan

REFERENCES:
- [Background] Fick DM, Cooper JW, Wade WE, Waller JL, Maclean JR, Beers MH. Updating the Beers criteria for potentially inappropriate medication use in older adults: results of a US consensus panel of experts. Arch Intern Med. 2003 Dec 8-22;163(22):2716-24. doi: 10.1001/archinte.163.22.2716. PMID 14662625
- [Background] Gallagher P, O'Mahony D. STOPP (Screening Tool of Older Persons' potentially inappropriate Prescriptions): application to acutely ill elderly patients and comparison with Beers' criteria. Age Ageing. 2008 Nov;37(6):673-9. doi: 10.1093/ageing/afn197. Epub 2008 Oct 1. PMID 18829684
- [Background] Krska J, Cromarty JA, Arris F, Jamieson D, Hansford D, Duffus PR, Downie G, Seymour DG. Pharmacist-led medication review in patients over 65: a randomized, controlled trial in primary care. Age Ageing. 2001 May;30(3):205-11. doi: 10.1093/ageing/30.3.205. PMID 11443021
- [Background] Laroche ML, Charmes JP, Merle L. Potentially inappropriate medications in the elderly: a French consensus panel list. Eur J Clin Pharmacol. 2007 Aug;63(8):725-31. doi: 10.1007/s00228-007-0324-2. Epub 2007 Jun 7. PMID 17554532